CLINICAL TRIAL: NCT02328521
Title: Efficacy Study of Nicorandil on Neointima After Coronary Drug-eluting Stent Implantation in Patients With Diabetic Mellitus
Brief Title: Efficacy Study of Nicorandil on Neointima
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhang Ying Qian (Other)
Responsible Party: Sponsor-Investigator, Zhang Ying Qian, M.D., Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2014-099-03; S2014-120-01 (Other: ChinaPLAGH)
Record Dates: First submitted 2014-12-24; First posted 2014-12-31 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Angina, Unstable; Diabetes Mellitus
Keywords: Neointima; Tomography, Optical Coherence; drug-eluting stents; Nicorandil
MeSH Terms: conditions — Angina, Unstable; Diabetes Mellitus; Neointima | interventions — Nicorandil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicorandil group (Experimental): Drug: Nicorandil (Chugai Pharmaceutical Co, Japan). The first dose is given 8h before selective percutaneous coronary intervention, 10mg, oral. After the percutaneous coronary intervention, nicorandil is given for 30 days, 5mg each time, 3 times daily oral.
  Interventions: Drug: Nicorandil
- Control group (Placebo Comparator): Drug: Nicorandil placebo (Sihuan Pharmaceutical Co, China). The first dose is given 8h before selective percutaneous coronary intervention, 2 tablets, oral. After the percutaneous coronary intervention, placebo is given for 30 days, 1 tablet each time, 3 times daily oral.
  Interventions: Drug: nicorandil placebo

INTERVENTIONS:
Drug: Nicorandil — Nicorandil is given once before PCI and given 3 times daily for 30 days after PCI.
  Other Names: Sigmart
  Arms: Nicorandil group
Drug: nicorandil placebo — Nicorandil placebo is given once before PCI and given 3 times daily for 30 days after PCI.
  Other Names: no other names
  Arms: Control group

SUMMARY:
The investigators aim to investigate the effect of oral nicorandil on neointima after coronary drug-eluting stent implantation in patients with diabetic mellitus.

DETAILED DESCRIPTION:
In the era of bare metal stent (BMS), the restenosis rate was about 25%. The introduction of drug-eluting stent (DES) reduces restenosis rate to 4%-10%. Neointimal hyperplasia and restenosis remain to be problems after DES implantation. Besides, DES causes an increase in uncovered struts, late stent thrombosis, neoatherosclerosis, and heterogeneous neointima. Diabetes mellitus (DM) results in increased risk for atherosclerosis, in-stent restenosis, neoatherosclerosis and late-stent thrombosis. Nicorandil, a hybrid of adenosine triphosphate-sensitive potassium (K-ATP) channel opener and nitrates, has been shown to reduce target vessel revascularization after stent implantation, target lesion revascularization after rotational atherectomy, and restenosis in patients undergoing percutaneous coronary intervention (PCI). Intracoronary optical coherence tomography(OCT) has emerged as a high-resolution imaging method for analysis of neointima that grows over the stent. We aim to examine the effect of nicorandil on the neointima after coronary DES implantation in patients with unstable angina and DM.

ELIGIBILITY:
Inclusion Criteria:

* unstable angina with diabetes mellitus and is not given glibenclamide
* have clinical indication of percutaneous coronary intervention
* de novo severe stenosis in a native coronary artery
* lesion suitable for stent and optical coherence tomography examination
* reference vessel size between 2.5 and 4.0mm
* drug-eluting stent implantation only

Exclusion Criteria:

* acute myocardial infarction within 2 weeks before percutaneous coronary intervention
* contraindications to treatment with nicorandil (allergy, glaucoma, digestive ulcer, is currently taking phosphodiesterase-5 inhibitor)
* bypass restenosis
* PCI history
* hypotension
* intolerance of platelet inhibitors and statins
* impaired liver function
* renal insufficiency requiring hemodialysis
* pregnancy
* connective tissue disease
* life expectancy ≤ 12 months
* left main coronary artery disease
* bypass graft lesion and lesions unsuitable for OCT
* unwillingness or inability to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Neointimal thickness (in μm) | 9 month
  Neointimal thickness is defined as the distance between the stent strut and lumen surface.
Neointimal area | 9 month
  Stent and lumen areas will be measured, and neointimal area is calculated as stent area minus lumen area.

SECONDARY OUTCOMES:
number of uncovered stent struts | 9 month
percent of uncovered stent struts | 9 month
characteristics of neointima (number of homogenous neointimal,number of layered neointima, number of heterogeneous neointima) | 9 month
  The characteristics of neointimal hyperplasia will be assessed and classified into three patterns according to the neointimal signal intensity.
number of in-stent neoatherosclerosis | 9 month
angiographic late lumen loss (in mm) | 9 month
  Late lumen loss is the difference of baseline and follow-up minimal luminal diameters.
rate of restenosis (in %) | 9 month
number of major adverse cardiovascular events | 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, M.D., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] IONA Study Group. Effect of nicorandil on coronary events in patients with stable angina: the Impact Of Nicorandil in Angina (IONA) randomised trial. Lancet. 2002 Apr 13;359(9314):1269-75. doi: 10.1016/S0140-6736(02)08265-X. PMID 11965271
- [Background] Horinaka S, Yabe A, Yagi H, Ishimitsu T, Yamazaki T, Suzuki S, Kohro T, Nagai R; JCAD Study Investigators. Effects of nicorandil on cardiovascular events in patients with coronary artery disease in the Japanese Coronary Artery Disease (JCAD) study. Circ J. 2010 Mar;74(3):503-9. doi: 10.1253/circj.cj-09-0649. Epub 2010 Jan 18. PMID 20081320
- [Background] Machecourt J, Danchin N, Lablanche JM, Fauvel JM, Bonnet JL, Marliere S, Foote A, Quesada JL, Eltchaninoff H, Vanzetto G; EVASTENT Investigators. Risk factors for stent thrombosis after implantation of sirolimus-eluting stents in diabetic and nondiabetic patients: the EVASTENT Matched-Cohort Registry. J Am Coll Cardiol. 2007 Aug 7;50(6):501-8. doi: 10.1016/j.jacc.2007.04.051. Epub 2007 Jul 23. PMID 17678732
- [Background] Kawai Y, Hisamatsu K, Matsubara H, Dan K, Akagi S, Miyaji K, Munemasa M, Fujimoto Y, Kusano KF, Ohe T. Intravenous administration of nicorandil immediately before percutaneous coronary intervention can prevent slow coronary flow phenomenon. Eur Heart J. 2009 Apr;30(7):765-72. doi: 10.1093/eurheartj/ehp077. Epub 2009 Mar 10. PMID 19276198
- [Background] Shehata M. Cardioprotective effects of oral nicorandil use in diabetic patients undergoing elective percutaneous coronary intervention. J Interv Cardiol. 2014 Oct;27(5):472-81. doi: 10.1111/joic.12142. Epub 2014 Aug 30. PMID 25174952
- [Background] Nagoshi R, Shinke T, Otake H, Shite J, Matsumoto D, Kawamori H, Nakagawa M, Kozuki A, Hariki H, Inoue T, Ohsue T, Taniguchi Y, Iwasaki M, Nishio R, Hiranuma N, Konishi A, Kinutani H, Miyoshi N, Takaya T, Yamada S, Yasaka Y, Hayashi T, Yokoyama M, Kato H, Kadotani M, Ohnishi Y, Hirata K. Qualitative and quantitative assessment of stent restenosis by optical coherence tomography: comparison between drug-eluting and bare-metal stents. Circ J. 2013;77(3):652-60. doi: 10.1253/circj.cj-12-0610. Epub 2012 Dec 21. PMID 23257388
- [Background] Tian F, Chen Y, Liu H, Zhang T, Guo J, Jin Q. Assessment of characteristics of neointimal hyperplasia after drug-eluting stent implantation in patients with diabetes mellitus: an optical coherence tomography analysis. Cardiology. 2014;128(1):34-40. doi: 10.1159/000357612. Epub 2014 Feb 7. PMID 24514877
- [Background] Chen J, Zhou S, Jin J, Tian F, Han Y, Wang J, Liu J, Chen Y. Chronic treatment with trimetazidine after discharge reduces the incidence of restenosis in patients who received coronary stent implantation: a 1-year prospective follow-up study. Int J Cardiol. 2014 Jul 1;174(3):634-9. doi: 10.1016/j.ijcard.2014.04.168. Epub 2014 Apr 21. PMID 24809921